CLINICAL TRIAL: NCT00708448
Title: Development of an Integrated Molecular Biomarker ofEarly Prediction of Therapeutic Response to Targeted Therapy in Stage IIIB/IV or Recurrent Lung Cancer Patients Using Imaging Assessments and Genomic Modeling
Brief Title: Early Prediction of Therapeutic Response to Targeted Therapy in Stage IIIB/IV or Recurrent Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI26198
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Radiation: PET Imaging; Drug: Erlotinib; Drug: Bevacizumab

INTERVENTIONS:
Radiation: PET Imaging — Patients will receive an FLT-PET scan, FDG-PET scan, a H215O-PET scan, and have a blood sample (15 cc, approximately 3 teaspoons) drawn for the genetic and protein studies. These studies will be done before patients begin taking erlotinib and bevacizumab.
  Other Names: FLT-PET scan, FDG-PET scan, a H215O-PET scan
Drug: Erlotinib — 150 mg/day
Drug: Bevacizumab — 15mg/kg q 21 days

SUMMARY:
This exploratory clinical study is designed to obtain pre-therapeutic imaging assessments using positron emission tomography (PET) imaging in 21 patients with Stage IIIB/IV or recurrent non-small cell lung cancer (NSCLC) and an early post therapy assessment at baseline and at various early time points (2 weeks in 7 patients, 4 weeks in 7 patients, and 6 weeks in 7 patients) after institution of erlotinib (anti-EGFR) (Tarceva) and bevacizumab (anti-VEGF) (Avastin) for first-line treatment of Stage IIIB/IV or recurrent non-squamous NSCLC. The proposed PET imaging and blood derived biomarkers trial is a companion study to an approved therapeutic trial (IRB# 24377). The therapeutic trial of erlotinib (Tarceva) and bevacizumab (Avastin) for first-line treatment of Stage IIIB/IV or recurrent lung cancer with drug costs exceeding $150,000 per patient/year (study drug budget exceeds $5 million) was funded for study at the HCI and the HICCP, statewide trial network. The proposed imaging study has been funded by the University of Utah Synergy Grant Program. The clinical imaging biomarkers will include an assessment of tumor metabolism [Banrasch 1986, Frauwirth 2002, Garber 2006, Kelloff 2005, Pauwels 1998, Semenza 2001, Smith 1999, Smith 2000, Sokoloff 1977, Warburg 1956, Weber 1977A, Weber] (dynamic FDG-PET); tumor proliferation [Rasey 2002,Shields 2001,Shields 1998, Vesselle 2002, Schwartz 2003] (dynamic FLT-PET); tumor blood flow and perfusion( H215O-PET)[Lodge 2000]; and tumor blood volume of distribution ( H215O -PET)[Lodge 2000] in the same patient at baseline and then in the same patient at one of the post therapy time points (2 weeks, 4 weeks, or 6 weeks). The investigators hypothesize that by using a set of imaging derived biomarkers and biomarkers from blood they can predict response, either prior to or at an earlier time point than would normally be determined with standard imaging techniques, in patients with lung cancer receiving combined bevacizumab and erlotinib.

DETAILED DESCRIPTION:
Non-Small Cell Lung Cancer Non- small cell lung cancer is the most common cause of cancer mortality in the United States [Jermal, 2007]. Surgery can be curative for patients with stages I and II disease and chemoradiation for curative intent can be administered to selected patients with stage III disease in the setting of adequate performance status, minimal comorbid disease and absence of weight loss. Adjuvant therapy improves survival, but the relapse rate is high and may approach 80% for subsets of patients with presumed "curable disease". Consequently, 85% of patients diagnosed with NSCLC will ultimately die of uncontrolled systemic disease. Systemic chemotherapy for treatment of metastatic disease, offers palliative benefit, improves survival, has substantial side effects, but is not curative. Improved systemic therapy with a greater therapeutic index due to greater efficacy or fewer side effects is sorely needed. Bevacizumab and/or erlotinib demonstrate these features.

Therapeutic Drugs (Erlotinib and Bevacizumab) The therapeutic trial, which this molecular imaging and serum biomarker trial will compliment, will study the combination of erlotinib and bevacizumab as first-line treatment for patients with non-squamous non-small cell lung cancer (NSCLC). This will be the first ever study where conventional chemotherapy will not be used as first-line treatment in NSCLC. Both erlotinib, as a single agent after chemotherapy progression [Shepherd 2005], and bevacizumab, in combination with chemotherapy [Sandler 2006], have been approved for the treatment of metastatic NSCLC. This is a multi-center trial via Huntsman Cancer Institute - Intermountain Cancer Care Program, phase II, single stage, of erlotinib (150 mg/day) and bevacizumab (15 mg/kg IV every 21 days) for patients with non-squamous, NSCLC without brain metastases or significant hemoptysis who have not received conventional chemotherapy as treatment for systemic or relapsed disease. Study treatment will be continued until symptomatic or objective progression. Patients progressing on or after this combination will subsequently receive conventional chemotherapy with bevacizumab at the discretion of the patient and treating physician. The study will be followed by the Data and Safety Monitoring Committee of the HCI and will enroll 40 patients. An interim safety analysis is scheduled after 20 patients have been accrued.

For purposes of defining response the following criteria are used for all target lesions: complete response-the disappearance of all target lesions; partial response-at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter; progressive disease-at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions; stable disease-neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.

The primary exploratory objectives of the study are:

* Provide a reliable and validated cadre of PET imaging derived biomarkers and serum derived biomarkers that yield a better understanding of: 1) early clinical benefit from Avastin and Tarceva therapy, 2) efficacy during Avastin and Tarceva therapy, and 3) prognosis or other long term outcomes.
* Reveal a more detailed understanding of: (1) the in vivo biologic mechanisms of Avastin and Tarceva in lung cancer and (2) information on why particular functional imaging assays and genomic biomarker profiles are seen in treated patients.
* Reveal a more detailed understanding of how the combination of molecular imaging derived biomarkers in combination with gene expression profiles/biomarkers will be potentially useful to physicians for decision making and for explanation of efficacy or outcomes for patients with cancer.
* Predict which patients may benefit from combined Avastin and Tarceva therapy.
* Determine early in the course of treatment whether Avastin and Tarceva will be efficacious and whether the imaging derived biomarkers in combination with blood derived biomarkers can be used in the future in patients with other types of malignancies to predict early response and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be enrolled in the the therapeutic trial (IRB # 24377) with non-squamous non-small cell lung cancer (NSCLC) treated with combined erlotinib (Tarceva) (150 mg/day)and bevacizumab (Avastin) (15mg/kg q 21 days) as first line therapy.
2. Adults must have radiological evidence of Stage IIIB/IV or recurrent non-squamous non-small cell carcinoma. The Stage IIIB/IV or Recurrent lesion must be in a location that includes a large arterial vessel to allow for determination of the H215O arterial input function. A previous histological diagnosis of NSCLC would be required prior to institution of therapy. Only clinically indicated biopsy and/or surgery for determination of Stage IIIB/IV or recurrent disease will be done and surgery is incidental to inclusion in the protocol.
3. Patients must be 18 years or older for inclusion in this study. Since there is no experience with [F-18]FLT in children and it would be inappropriate to study individuals under the age of 18 until more safety data is available.
4. After entry into the study, patients are expected to be followed for at least 2 months as part of standard of care.
5. All patients, or their legal guardians, must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
6. The patient, if female, must be postmenopausal for a minimum of one year or surgically sterile, or on one of the following methods of birth control for a minimum of one month prior to entry into this study: IUD, oral contraceptives, Depo-Provera or Norplant. These criteria can be waived at the discretion of the investigator if the patient's tumor is considered life threatening and the one month wait required is not in the best interest of the patient. Negative pregnancy test is accepted.
7. Pre-treatment laboratory tests for patients receiving [F-18]FLT must be performed within 21 days prior to study entry. These must be less than 4 times below or above the upper or lower limit range for the respective laboratory test. The patients have Stage IIIB/IV or recurrent NSCLC and therefore many routine laboratory tests may not be within the typical normal range. Using a factor of 4 times above or below the upper or lower value for the normal range for laboratory test will assure ability to recruit patients and maintain safety. In those instances where a value of 4X above the normal range would be inappropriate for inclusion (prothrombin time and partial thromboplastin time) then a value of 2.5X will be used for these two laboratory tests. In those instances when the prothrombin time or partial thromboplastin time are greater than 2.5X the upper limit of normal then such a patient would not be enrolled. The 4X value will be used for all laboratory values except prothrombin time and partial thromboplastin time which cannot be above or below 2.5 times the upper or lower limit of normal (Appendix E, [F-18]FLT Laboratory Study Results). A negative serum pregnancy test is required within 2 days prior to the PET studies.
8. Pre-treatment radiological clinical scans/studies (Gd- enhanced MRI or CT to document Stage IIIB/IV or recurrent NSCLC) must be performed within 30 days of study entry.

Exclusion Criteria:

1. Patients will be receiving erlotinib (Tarceva) (150 mg/day)and bevacizumab (Avastin) (15mg/kg q 21 days) as part of the therapeutic trial. Enrollment may not occur if the patient does not meet the enrollment criteria for the therapeutic trial
2. Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
3. Patients who are pregnant or lactating or who suspect they might be pregnant.
4. Adult patients who require monitored anesthesia for PET scanning.
5. HIV positive patients due to the previous toxicity noted with FLT.
6. Claustrophobia or inability to remain stationary within the PET scanner for 90 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03-28 (Actual); Primary Completion 2010-08-12 (Actual); Study Completion 2010-08-12 (Actual)

PRIMARY OUTCOMES:
Provide reliable validated, PET imaging derived biomarkers and serum derived biomarkers for a better understanding of early clinical benefit from Avastin/Tarceva therapy, efficacy during Avastin/Tarceva therapy, and prognosis or other long term outcomes. | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- See also: NCT00585377 (Companion Protocol) — http://clinicaltrials.gov/ct2/show/NCT00585377?term=Akerley&rank=2